CLINICAL TRIAL: NCT04371783
Title: A Randomized Trial Comparing the Live Birth Rate of Immediate Versus Delayed Frozen Embryo Transfer (FET) Replacing a Single Blastocyst in the First FET of the First Stimulated IVF Cycle Following a Freeze-all Strategy
Brief Title: A Randomized Trial Comparing the Live Birth Rate of Immediate Versus Delayed FET Following a Freeze-all Strategy
Acronym: FET
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ShangHai Ji Ai Genetics & IVF Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JIAI 2020-04
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-05

CONDITIONS: IVF; Frozen Embryo Transfer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate FET group (Other): FET will be performed in the first menstrual cycle following the stimulated IVF cycle
  Interventions: Procedure: Immediate FET
- Delayed FET group (Other): FET will be performed in the second menstrual cycle following the stimulated IVF cycle
  Interventions: Procedure: Delayed FET

INTERVENTIONS:
Procedure: Immediate FET — FET is performed in the first menstrual cycle following the stimulated IVF cycle
  Arms: Immediate FET group
Procedure: Delayed FET — FET is performed in the second menstrual cycle following the stimulated IVF cycle
  Arms: Delayed FET group

SUMMARY:
This randomized trial we aim to compare the live birth rate of immediate versus delayed FET replacing a single blastocyst in the first FET of the first stimulated IVF cycle following. The hypothesis is that the live birth rate of the immediate FET is higher than the delayed FET replacing a single blastocyst in the first FET of the first stimulated IVF cycle following a freeze-all strategy. Women will undergo IVF/ICSI in the centre as clinically indicated. Standard ovarian stimulation with gonadotrophins in a Gonadotrophin releasing hormone (GnRH) antagonist protocol will be employed. Hormone replacement treatment (HRT) will be used in subsequent FET cycles. On Day 3 of the menstrual cycle, we will measure the anxiety levels using the Chinese State-Trait Anxiety Inventory and serum E2, cortisol levels will be checked on the same day.

Recruited women having the first FET cycle following a freeze all strategy will be randomly assigned on the day of blastocyst(s) freezing according to a computer-generated randomization list into one of the following two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 20-40 years at the time of IVF/ICSI
2. Women undergoing their first FET of the first IVF cycle following a freeze-all strategy
3. Undergoing IVF with GnRH antagonist
4. At least one frozen blastocyst

Exclusion Criteria:

1. Severe ovarian hyperstimulation syndrome during the first IVF/ICSI cycle
2. Preimplantation genetic testing
3. Use of donor oocytes
4. Presence of untreated hydrosalpinx or endometrial polyp on scanning during ovarian stimulation

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 828 (Estimated)
Dates: Start 2020-05-04 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
live birth | 1 year after FET
  deliveries ≥22 weeks gestation with heartbeat and breath

SECONDARY OUTCOMES:
positive hCG | 2 weeks after FET
  serum β-hCG ≥10 mIU/mL
clinical pregnancy | 6 weeks' gestation
  presence of intrauterine gestational sac by trans-vaginal ultrasound at 6 gestational weeks.
ongoing pregnancy | 12 weeks' gestation
  a viable pregnancy beyond 12 weeks' gestation
implantation rate | 6 weeks' gestation
  the number of gestational sacs per blastocyst transferred
miscarriage | 1 year after FET
  a clinically recognized pregnancy loss before the 22 weeks of pregnancy
multiple pregnancy | multiple pregnancy beyond gestation 12 weeks
  more than one intrauterine sacs on scanning
ectopic pregnancy | ectopic pregnancy during 12 weeks gestation
  pregnancy outside the uterine cavity
birthweight of newborns | 1 year after FET
  the birth weight of newborns

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxi Sun, Phd, Study Director — Shanghai JiAi Genetics & IVF Institute
Locations (1):
- Shanghai JiAi Genetics & IVF Institute, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results after deidentification (text, tables, figures, and appendices) and study protocol will be shared.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will be available when beginning 3 months and ending 5 years following article publication.
Access Criteria: To achieve aims in the approved proposal, researchers who provide a methodologically sound proposal will be shared with. Proposals should be directed to lihe198900@163.com.

REFERENCES:
- [Background] Doody KJ. Cryopreservation and delayed embryo transfer-assisted reproductive technology registry and reporting implications. Fertil Steril. 2014 Jul;102(1):27-31. doi: 10.1016/j.fertnstert.2014.04.048. Epub 2014 Jun 4. PMID 24907917
- [Background] Shapiro BS, Daneshmand ST, Garner FC, Aguirre M, Hudson C, Thomas S. Evidence of impaired endometrial receptivity after ovarian stimulation for in vitro fertilization: a prospective randomized trial comparing fresh and frozen-thawed embryo transfer in normal responders. Fertil Steril. 2011 Aug;96(2):344-8. doi: 10.1016/j.fertnstert.2011.05.050. Epub 2011 Jul 6. PMID 21737072
- [Background] Venetis CA, Kolibianakis EM, Bosdou JK, Lainas GT, Sfontouris IA, Tarlatzis BC, Lainas TG. Estimating the net effect of progesterone elevation on the day of hCG on live birth rates after IVF: a cohort analysis of 3296 IVF cycles. Hum Reprod. 2015 Mar;30(3):684-91. doi: 10.1093/humrep/deu362. Epub 2015 Jan 12. PMID 25586787
- [Background] Santos-Ribeiro S, Polyzos NP, Lan VT, Siffain J, Mackens S, Van Landuyt L, Tournaye H, Blockeel C. The effect of an immediate frozen embryo transfer following a freeze-all protocol: a retrospective analysis from two centres. Hum Reprod. 2016 Nov;31(11):2541-2548. doi: 10.1093/humrep/dew194. Epub 2016 Sep 8. PMID 27609984
- [Background] Santos-Ribeiro S, Siffain J, Polyzos NP, van de Vijver A, van Landuyt L, Stoop D, Tournaye H, Blockeel C. To delay or not to delay a frozen embryo transfer after a failed fresh embryo transfer attempt? Fertil Steril. 2016 May;105(5):1202-1207.e1. doi: 10.1016/j.fertnstert.2015.12.140. Epub 2016 Jan 21. PMID 26806686
- [Background] Lattes K, Checa MA, Vassena R, Brassesco M, Vernaeve V. There is no evidence that the time from egg retrieval to embryo transfer affects live birth rates in a freeze-all strategy. Hum Reprod. 2017 Feb;32(2):368-374. doi: 10.1093/humrep/dew306. Epub 2016 Dec 16. PMID 27986819
- [Background] Volodarsky-Perel A, Eldar-Geva T, Holzer HE, Schonberger O, Reichman O, Gal M. Cryopreserved embryo transfer: adjacent or non-adjacent to failed fresh long GnRH-agonist protocol IVF cycle. Reprod Biomed Online. 2017 Mar;34(3):267-273. doi: 10.1016/j.rbmo.2016.11.013. Epub 2016 Dec 16. PMID 28041829
- [Background] Higgins C, Healey M, Jatkar S, Vollenhoven B. Interval between IVF stimulation cycle and frozen embryo transfer: Is there a benefit to a delay between cycles? Aust N Z J Obstet Gynaecol. 2018 Apr;58(2):217-221. doi: 10.1111/ajo.12696. Epub 2017 Sep 14. PMID 28905357
- [Derived] Li H, Zhang W, Chen J, Lu X, Li L, Sun X, Ng EH. Immediate versus delayed single blastocyst transfer following the first stimulated IVF cycle in the freeze-all strategy: a study protocol for a randomised controlled trial. BMJ Open. 2024 May 8;14(5):e081018. doi: 10.1136/bmjopen-2023-081018. PMID 38719320